CLINICAL TRIAL: NCT04240119
Title: Angiogenic Factors in Stroke (ANFIS)
Brief Title: Angiogenic Markers in Cerebrovascular Disease (ANFIS)
Acronym: ANFIS
Status: Enrolling by invitation | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Nestor R. Gonzalez, MD, MSCR., Professor of Neurosurgery, Cedars-Sinai Medical Center
Other Study IDs: Pro00046030
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Transient Ischemic Attack; Atherosclerosis; Intracranial Arterial Stenosis; Moyamoya
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Atherosclerosis; Moyamoya Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: According to current clinical care standards — Enrolled subjects may be treated with medical management or surgically using indirect revascularization surgery.

SUMMARY:
Intracranial atherosclerosis (ICAS) is the most common cause of stroke worldwide. It carries a worse prognosis than other stroke etiologies, with an annual rate of recurrent stroke and death of 15% despite intensive medical management, and as high as 35% in certain populations. Overall, treatment and prevention of stroke due to ICAS has been unsuccessful. While two recent clinical trials have shown modest improvement in the efficacy of intensive medical treatment, these trials were terminated early given the elevated rate of complications, stroke, and death in the interventional arms. In fact, intensive medical management appears to reduce the risk of embolism; however, medical management alone does not address the progression of intracranial arterial stenosis or the pathophysiologic components of hypoperfusion and poor collateral circulation.

Levels and types of various angiogenic factors in the blood and tissues have been proposed to be predictive of patient outcome after ischemic stroke and treatment for stroke. This study therefore pursues a new paradigm to investigate responses to ICAS treatment from the perspective of cerebral collateral vessel generation and the role of angiogenic factors. Specifically, pro- and anti-angiogenic factors in patients with ICAS are evaluated at baseline and longitudinally in response to both medical and surgical treatment. For this we have developed methodologies for the isolation and measurement of these growth factors in plasma of patients with ICAS. These methodologies will enable us to obtain a detailed understanding of the variation and dynamic properties of local and circulating angiogenic factors over time in response to medical and surgical treatment, and their association to outcome phenotypes. This analysis is complemented by studies of angiographic development of neovascularization. If successful, this study will help to better understand the role of angiogenesis in ICAS and create a foundation from which to explore therapeutic treatments for ICAS which harness the natural processes of angiogenesis.

DETAILED DESCRIPTION:
Intracranial atherosclerosis (ICAS) is the most common cause of stroke worldwide. It accounts for at least 10% of all strokes in the United States and as much as 67% in countries with predominantly Asian, Hispanic, and Black populations. ICAS carries a worse prognosis than other stroke etiologies, with an annual rate of recurrent stroke and death of 15% despite intensive medical management, and as high as 35% in certain populations. Recent randomized controlled clinical trials have shown that angioplasty with stenting and bypass surgery fail to improve outcomes in patients with ICAS.

Overall treatment and prevention of stroke due to ICAS has been unsuccessful. The results of two recent clinical trials exploring interventions for the management of cerebrovascular occlusive disease-bypass surgery (Carotid Occlusion Surgery Study [COSS]) and angioplasty and stenting (SAMMPRIS)-have shown modest improvement in the efficacy of intensive medical treatment. However, both trials were terminated early given the elevated rate of complications, stroke, and death in the interventional arms. In the medical arms of COSS and SAMMPRIS, the rates of stroke and death at two years were 21% and 15%, respectively. Intensive medical management appears to reduce the risk of embolism; however, medical management alone does not address the progression of intracranial arterial stenosis or the pathophysiologic components of hypoperfusion and poor collateral circulation. Patients with prior stroke had an even higher rate of stroke, 35%.

Levels and types of various angiogenic factors in the blood and tissues have been proposed to be predictive of patient outcome after ischemic stroke and treatment for stroke. This study therefore pursues a new paradigm to investigate responses to ICAS treatment from the perspective of cerebral collateral vessel generation and the role of angiogenic factors. Specifically, pro- and anti-angiogenic factors in patients with ICAS are evaluated at baseline and longitudinally in response to both medical and surgical treatment. For this we have developed methodologies for the isolation and measurement of these growth factors in plasma of patients with ICAS. These methodologies will enable us to obtain a detailed understanding of the variation and dynamic properties of local and circulating angiogenic factors over time in response to medical and surgical treatment, and their association to outcome phenotypes. This analysis is complemented by studies of angiographic development of neovascularization. If successful, this study will help to better understand the role of angiogenesis in ICAS and create a foundation from which to explore therapeutic treatments for ICAS which harness the natural processes of angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* 70% to 99% ICAS of a major intracranial artery diagnosed by angio, TCD, MRA, or CTA.

Exclusion Criteria:

* Intracranial tumor or vascular malformation.
* Any hemorrhagic infarct within 14 days before enrollment or any other intracranial hemorrhage (subarachnoid, subdural, or epidural) within 30 days.
* Intracranial arterial stenosis related to arterial dissection or any known infectious or vasculitic disease.
* Presence of any unequivocal cardiac sources of embolism.
* Major surgery within previous 30 days before enrollment or planned in the next 180 days after enrollment,
* Severe neurologic deficit that renders the patient incapable of living independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during hospitalizations or neurological and/or neurosurgical office visits at Cedars Sinai Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-07; Primary Completion 2030-07 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurring cerebrovascular events | 2 years
Plasma levels of angiogenic factors | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nestor R Gonzalez, MD., MSCR, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared in the future, but currently no specific plans exist.